CLINICAL TRIAL: NCT04231812
Title: First In Human Study Evaluating the Safety and Performance of the "LapBox" Containment System for Laparoscopic Tissue Morcellation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ARKSurgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ARK-001
Record Dates: First submitted 2019-12-24; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Laparoscopic Surgical Procedure
Keywords: Laparoscopic Tissue Morcellation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- open lable (Other): Prospective, open-label
  Interventions: Device: Laparoscopic Tissue Morcellation working space (bag)

INTERVENTIONS:
Device: Laparoscopic Tissue Morcellation working space (bag) — The "LapBox" is working space (bag) intended for use as a laparoscopic instrument port and tissue containment system that creates a working space allowing for visualization during power or manual morcellation procedure following a laparoscopic procedure for the excision of benign gynecologic tissue that is not suspected to contain malignancy

SUMMARY:
Study to assess the safety, and performance of the LapBox in patients in terms of duration of deployment, organ insertion into the "LapBox" bag, ease of use, success of containment and performance.

DETAILED DESCRIPTION:
The LapBox is intended for use as a laparoscopic instrument port and tissue containment system that creates a working space allowing for visualization during power or manual morcellation procedure following a laparoscopic procedure for the excision of benign gynecologic tissue that is not suspected to contain malignancy Ten (10) adult female patients, scheduled for the laparoscopic gynecological procedure, with up to 700gr mass to be removed and with no suspicion of malignancy.

Patients scheduled for elective laparoscopic hysterectomy, myomectomy or removal of an adnexal mass where either manual morcellation or power morcellation is needed for tissue will be enrolled. Each patient will be required to participate in 3 visits:

Visit 1: Screening and Enrollment, as part of the pre-operative visit and confirmation of compliance. Such a visit can be more than 1 day.

Visit 2: Laparoscopic organ removal procedure- morcellation utilizing LapBox containment system.

Visit 3:up appointment up to 7 weeks (7 days) post-procedure.

During visit 2 (laparoscopic organ removal procedure), the following steps will be performed:

* Following tissue harvest and prior to morcellation, a peritoneal wash sample will be obtained for a cytology evaluation.
* The LapBox will then be inserted to the patient abdomen through the abdominal wall and deployed.
* The harvested tissue will be inserted into the LapBox using standard technique.
* The LapBox opening will be extracted outside the abdomen.
* Depending on the type of morcellation (power or mechanical), the incision may be extended as needed.
* The appropriate type of port will be placed.

Power morcellation:

* The morcellator will be inserted.
* The laparoscope will be placed inside the bag and provide visualization of the procedure. Alternatively, direct visualization may be utilized.
* The morcellator will be operated in a standardized fashion. Manual morcellation will be performed as per standard practice.
* The LapBox will be removed through the abdominal opening. A second peritoneal wash sample will be obtained for a cytology evaluation in order to compare pre and post morcellation findings.

Following the procedure, tissue weight will be recorded, and leakage testing will be performed on used devices.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients indicated for elective surgery requiring laparoscopic hysterectomy, myomectomy where either manual morcellation or power morcellation is needed for tissue removal at which a morcellator for cutting and extraction of tissue is required.
2. Pre- menopausal woman patient age 18-50 years
3. Mass measured with diameter up to 10 cm to be removed
4. Normal Pap test result within the last 24 months prior to enrollment
5. Normal and /or Non-Clinically Significant as per investigator discretion CBC and Blood chemistry test within at least 6 months prior to surgery.
6. Signed an informed consent

Exclusion Criteria:

1. Emergency cases
2. Abdominal wall thickness is greater than 10 cm according to US measurements.
3. Patient requires procedure involving the ovaries (e.g., Oophorectomy, Salpingo)
4. Patient is defined as a "high risk" patient for developing cancer (per standard assessment, including but not limited to imaging)
5. Suspicion of malignant or pre-malignant tissue according to preoperative assessment including US exam within 30 days prior to surgery
6. Known or suspected gynecologic malignancy within the past five years
7. Pacemaker, internal defibrillator/cardio converter
8. Previous extensive pelvic surgery or any other medical procedure which in the investigator's judgment contraindicates the patient's participation
9. Contraindications to anesthesia or abdominal surgery. ASA score above 3
10. Concurrent participation in any other clinical study
11. Active infection at the time of the procedure.
12. BMI<20 or BMI>40
13. Known history or presence of any medical disorder, which in the investigator's judgment contraindicates the patient's participation (e.g., Known and documented active liver disease, renal failure, cognitive disorder, cardiopulmonary disease, impaired coagulation parameters, etc.)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Intended use of the device -during the laparoscopic procedure for the excision of benign gynecologic tissue that is not suspected to contain malignancy
Enrollment: 10 (Estimated)
Dates: Start 2020-01-25 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Device Related Adverse Events Occurrence | through study procedure, up to 10 weeks from procedure
  Occurrence of device use related adverse events as documented and reported, under DSMB review
Device Performance and Integrity | following completion of procedure and study device use (1 day)
  Leak testing will be performed following the each procedure to confirm device integrity.
  Used device will be filled with color fluid to provide clear identification of possible leakage. Test will performed by Investigator delegated study team member and results will be documented in CRF.

SECONDARY OUTCOMES:
Device performance | up to 10 weeks following the procedure
  Comparison of the presence of cancerous cells pre and post morcellation via peritoneal wash sample cytology
Device Performance (usability) | following completion of procedure and study devise use (1 day)
  Ease of use of the device (usability evaluation via questionnaire).
Device Performance | through study procedure, up to 10 weeks from procedure
  Intra- or post-operative complications, Adverse Events and Device Related Adverse Events
Device Performance | following completion of procedure and study device use (1 day)
  Procedure time
Device Performance | up to 10 weeks following the procedure
  Hospitalization length
Device Performance | following completion of procedure and study devise use (1 day)
  Specimen (removed tissue) weight collection

CONTACTS AND LOCATIONS:
Overall Officials: Roy Mashiach, Dr, Principal Investigator — Assuta Tel Aviv Medical Center, Tel Aviv, Israel; Yuval Kaufman, Dr, Principal Investigator — Assuta Haifa Medical Center, Haifa, Israel